CLINICAL TRIAL: NCT00683826
Title: Effects of Leucine Supplement on Body Weight and Cardiometabolic Changes
Brief Title: The Effects of Leucine on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Henry N. Ginsberg, Herbert and Florence Irving Professor of Medicine; Director - Irving Institute for Clinical & Translational Research, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAC6762
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Overweight; Obesity
Keywords: Leucine; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- L-Leucine 4grams (Experimental): This will be a triple arm design where subjects will be randomized into three groups. Arm #1 will be 4g of Leucine.
  Interventions: Other: Liquid meal; Dietary Supplement: L-Leucine 4g
- L-Leucine 8 grams (Experimental): Arm number two of the study will be a dose of Leucine of 8g.
  Interventions: Dietary Supplement: L-Leucine 8gr; Other: Liquid meal
- L-Leucine 0 grams (Placebo Comparator): The third arm of the study will be composed of a control drink with no leucine in it.
  Interventions: Other: Liquid meal

INTERVENTIONS:
Dietary Supplement: L-Leucine 8gr — Supplementation in the form of a liquid meal (premixed leucine powder solutions with flavor made by the Bionutrition Unit of the Irving Insitute for Clinical and Translational Research (IICTR)). Dosing of leucine will be a combination of 2 ounces of liquid per 1 gm of leucine. L-leucine was purchased (FCC quality) from Spectrum Chemical,California. Certificate of analysis enclosed (99.89% leucine).Liquid meal preparation: Grape juice and crystal light mixes will be used for the preparation of liquid meals that will be given to each participant each week. Participants will consume two 8 ounce drinks (packaged in two 10 ounce bottles) per day. Each drink will be individually prepared with 8 grams of leucine.
  Arms: L-Leucine 8 grams
Other: Liquid meal — Liquid meal preparation (contents): Grape juice and crystal light mixes will be used for the preparation of liquid meals that will be given to each participant each week. Participants will consume two 8 ounce drinks (packaged in two 10 ounce bottles) per day. The placebo group will have the same drinks listed above with no leucine incorporated.
Dietary Supplement: L-Leucine 4g — Supplementation in the form of a liquid meal (premixed leucine powder solutions with flavor made by the Bionutrition Unit of the Irving Insitute for Clinical and Translational Research (IICTR)). Dosing of leucine will be a combination of 2 ounces of liquid per 1 gm of leucine. L-leucine was purchased (FCC quality) from Spectrum Chemical,California. Certificate of analysis enclosed (99.89% leucine).Liquid meal preparation: Grape juice and crystal light mixes will be used for the preparation of liquid meals that will be given to each participant each week. Participants will consume two 8 ounce drinks (packaged in two 10 ounce bottles) per day. Each drink will be individually prepared with 4 grams of leucine.
  Arms: L-Leucine 4grams

SUMMARY:
Protein-rich diets appear to show some benefits in promoting weight loss. It is thought that increased intake of leucine may account for some of this effect. This study is designed to assess whether any of the beneficial effects of dietary leucine supplementation observed in mice also apply to humans.

Specifically, our team would like to determine whether oral leucine supplementation in overweight/obese humans increases metabolic rate, reduces body weight, improves glucose utilization and/or, reduces circulating fat levels in the blood. We hope that the results obtained from this pilot study will highlight the specific aspects of metabolic improvement associated with increased daily leucine intake. This study will should provide data that can be used to design more definitive trials with regard to dietary leucine supplementation.

Hypothesis

This pilot study is designed to accomplish the following two goals:

1. to assess whether any of the beneficial effects of dietary leucine supplementation observed in mice also apply in humans. Specifically, we want to determine whether oral leucine supplementation in overweight/obese individuals' increases basal metabolic rate, reduces body weight, improves glucose tolerance and/or insulin sensitivity, and/or reduces circulating Low-density Lipoprotein (LDL)-cholesterol levels.
2. To provide data that can be used to design more definitive trials with regard to dietary leucine supplementation.

We hope that the results obtained from this pilot study will highlight the specific aspects of metabolic improvement associated with increased daily leucine intake. This would in turn lead to more rigorous clinical trials involving larger sample sizes, and with diverse populations of different gender, age, and ethnic groups. Future trials may also be directed to determine minimal doses and durations of leucine supplementation that are capable of achieving clinically significant improvement in the cardio-metabolic risk profile in people.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year old overweight/obese
* healthy men and women
* Body Mass Index (BMI) of 28-35

Exclusion Criteria:

* unusual or extreme dietary or exercise habits
* daily leucine supplement use
* inability to follow instructions to drink liquid meals
* type 1 diabetes or type 2 diabetes on drug treatment(diet controlled diabetics will be enrolled after consulting with their treating physicians)
* hypothyroidism or hyperthyroidism
* chronic wasting diseases (Acquired Immune Deficiency Syndrome (AIDS), cancers, cirrhosis, renal failure, Chronic Obstructive Pulmonary Disease (COPD), heart failure)
* drug or alcohol abuse
* tobacco smoker within the past 6 months
* pregnancy or lactating
* use of medications known to affect carbohydrate or lipid metabolism, satiety, or hunger
* anemia
* abnormal liver function tests (LFTs)
* women who are of child bearing age without adequate birth control modality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ginsberg, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was completed. All subjects were recruited from the surrounding neighborhood and affiliates of Columbia University Medical Center (CUMC).
Groups:
- All Study Participants: This will be a three-way crossover design, where subjects will be randomized into three groups. All subjects will receive all interventions (0g leucine, 4g leucine, 8g leucine) in a randomized order.
Period: Overall Study
Arm/Group | All Study Participants
Started | 8
0g Leucine | 8
8g Leucine | 8
4g Leucine | 7
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Leucine 4 Grams; Leucine 8 Grams; Leucine 0 Grams-control: Initial intervention.
- Total: Total of all reporting groups
Arm/Group | Leucine 4 Grams | Leucine 8 Grams | Leucine 0 Grams-control | Total
Number analyzed (Participants) | 2 | 3 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 8
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (7) | 40 (7) | 45 (7) | 40 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 7
  Male | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Effects on Weight
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Leucine 4 Grams: This will be a triple arm design where subjects will be randomized into three groups. Arm #1 will be 4g of Leucine.
- Leucine 8 Grams: Arm number two of the study will be a dose of Leucine of 8g.
- Leucine 0 Grams-control: The third arm of the study will be composed of a control drink with no leucine in it.
Arm/Group | Leucine 4 Grams | Leucine 8 Grams | Leucine 0 Grams-control
Number analyzed (Participants) | 7 | 8 | 8
kilograms | 93.4 (16.8) | 91.7 (17.2) | 91.9 (15.2)

2. Secondary Outcome: Energy Expenditure
Time Frame: will be measure at the end of each treatment period (6 weeks)
Reporting Status: Not Posted

3. Primary Outcome: Weight
Time Frame: at the end of each study treatment arm (six weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Leucine 4 Grams | Leucine 8 Grams | Leucine 0 Grams-control
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No